CLINICAL TRIAL: NCT00909298
Title: A Randomized Clinical Trial of Intrinsic Pathway Antagonists in Patients Undergoing Implantation of Left Ventricular Assist Devices
Brief Title: Left Ventricular Assist Device (LVAD) Specialized Centers of Clinically Orientated Research (SCCOR) Coagulation - Acute Intrinsic Pathway Antagonist (IPA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: vTv Therapeutics (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Alan Moskowitz, MD Co-Director, International Center for Health Outcomes and Innovation Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TTP889-202
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Coagulation
Keywords: Left ventricular assist devices; Cardiac Disease; Heart Failure; Anticoagulant for Left Ventricular Assist Devices
MeSH Terms: conditions — Thrombosis; Heart Diseases; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): TTP889 300 mg
  Interventions: Drug: TTP889
- 2 (Placebo Comparator): TTP889 Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TTP889 — 300 mg
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine if post-operative administration of intrinsic pathway antagonist (TTP889) in patients on Left Ventricular Assist Device (LVAD) support will result in a 50% reduction of thrombin generation markers at 28 days compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, release of medical information, and HIPAA forms
* Age greater than or equal to 18 years
* Male, postmenopausal female, or female who may become pregnant but is using adequate contraceptive precautions (defined as oral contraceptive, intrauterine devices, surgical contraception or a combination of a condom and a spermicide), with negative pregnancy test
* Implanted with an FDA-approved LVAD (for BTT or DT indication, e.g. HeartMate® XVE) within 72 hours prior to randomization, and able to receive the first dose of study drug by 72 hours (+6 hours) post LVAD implantation
* Post-op hemostasis adequate for starting low level anticoagulation (as assessed by surgeon)
* Extubated and able to take oral medication

Exclusion Criteria:

* Evidence of active bleeding within 24 hours prior to randomization
* History of a platelet disorder, including but not limited to thrombocytopenia and thrombasthenia
* Thrombocytopenia with platelets <80,000/ml within 48 hours prior to randomization
* History of an inherited or acquired coagulation disorder
* Hemoglobin <8 g/dL (4.85 mmol/L) or hematocrit <26% within 24 hours prior to randomization
* Clinical indication for (or the intention to use) standard anticoagulation therapy at time of randomization (e.g., atrial fibrillation or DVT)
* Intention to treat with more than 325 mg aspirin daily
* Any clinical requirement or intention to treat with phenytoin, tolbutamide or warfarin post randomization
* RVAD support at the time of randomization
* Estimated glomerular filtration rate (GFR) ≤30 ml/min (by Cockcroft-Gault formula), or any form of dialysis within 48 hours prior to randomization
* Evidence of intrinsic hepatic disease as defined as biopsy proven liver cirrhosis; or liver enzyme values (AST or ALT) that are >3 times the upper limit of normal; or Total Bilirubin >1.5 times the upper limit of normal (with the exception of Gilbert's Syndrome) within 3 days prior to randomization
* Active systemic infection, in the judgment of the investigator, within 3 days prior to randomization
* Stroke or transient ischemic attack (TIA) within 6 months prior to randomization
* History of intracranial hemorrhage or gastrointestinal bleed within 3 months prior to randomization
* Alzheimer's disease, or any other form of irreversible dementia
* History of psychiatric disease (including drug or alcohol abuse) that may impair compliance with the study protocol
* Pregnant or breastfeeding at time of randomization
* Received investigational intervention within 30 days prior to randomization
* Body weight < 45 Kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The level of thrombin generation markers | 28 days following initiation of study drug
  Thrombin-antithrombin complex (TAT)and Prothrombin Fragment 1+2 (F1.2)

SECONDARY OUTCOMES:
Thrombin Generation Markers | Baseline, Days 1, 3, 5, 7, 14, 21, 28 (±2); and 42 (± 4) days post-randomization
Major Bleeding | Day 1 to Day 42 (± 4) days post-randomization
Transfusions of Blood and Blood Products | Days 1, 3, 5, 7, 14, 21, 28 (±2); and 42 (± 4) days post-randomization
Blood Count | Baseline, Days 1, 3, 5, 7, 14, 21, 28 (±2); and 42 (± 4) days post-randomization
Coagulation Markers | Baseline, Days 1, 3, 5, 7, 14, 21, 28 (±2); and 42 (± 4) days post-randomization
Incidence of Serious Adverse Events | Baseline, Days 1, 3, 5, 7, 14, 21, 28 (±2); and 42 (± 4) days post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Alan Moskowitz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Yoshifumi Naka, MD, PhD, Principal Investigator — New York Presbyterian Hospital / Columbia University Medical Center
Locations (3):
- United States (3):
  - Mount Sinai School of Medicine, New York, New York
  - New York Presbyterian Hospital / Columbia University Medical Center, New York, New York
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington